CLINICAL TRIAL: NCT00281528
Title: A Phase II Study of Weekly Versus Every 2-week Versus Every 3-week Administration of ABI-007 (Abraxane) in Combination With Bevacizumab in Women With Metastatic Breast Cancer.
Brief Title: Weekly vs. Every 2 Week vs. Every 3 Week Administration of ABI-007 (Abraxane)/Bevacizumab Combination in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sufficient mature data to complete a final analysis
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA023
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2012-03-13 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: First Line Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 260 mg/m^2 ABI-007 every 3 weeks (Experimental): 260 mg/m^2 every 3 weeks and 15 mg/kg bevacizumab every 3 weeks
  Interventions: Drug: ABI-007 (Abraxane); Drug: bevacizumab
- 260 mg/m^2 ABI-007 every 2 weeks (Experimental): 260 mg/m^2 ABI-007 every 2 weeks and 10 mg/kg bevacizumab every 2 weeks
  Interventions: Drug: ABI-007 (Abraxane); Drug: bevacizumab
- 130 mg/m^2 ABI-007 weekly (Experimental): 130 mg/m^2 ABI-007 weekly (without a week of 'rest') and 10 mg/kg bevacizumab every 2 weeks
  Interventions: Drug: ABI-007 (Abraxane); Drug: bevacizumab

INTERVENTIONS:
Drug: ABI-007 (Abraxane) — 30 minute infusions
  Other Names: Abraxane; paclitaxel bound to albumin
Drug: bevacizumab — infusions
  Other Names: Avastin

SUMMARY:
This is a multi-center, open-label, randomized Phase II study in previously untreated patients with metastatic breast cancer to evaluate the antitumor activity and safety of weekly dose-dense ABI-007 (Abraxane) compared to 2-weekly regimen vs the standard 3-weekly infusion. All patients will also receive concurrent bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the breast.
* Stage IV disease
* Measurable disease
* Patients must not be a candidate for Herceptin therapy
* At least 4 weeks since radiotherapy, with full recovery. The measurable disease must be completely outside the radiation portal or there must be pathologic proof of progressive disease within the radiation portal.
* At least 4 weeks since major surgery, with full recovery.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Female >18 years of age.
* Patient has the following blood counts at Baseline:

Absolute neutrophil count ≥ 1.5 x 10^9cells/L; platelets ≥ 100 x 10^9 cells/L; hemoglobin ≥ 9 g/dL.

* Patient has the following blood chemistry levels at Baseline: Aspartate transaminase (AST or SGOT), alanine aminotransferase (ALT or SGPT) ≤ 2.5x upper limit of normal range (ULN); total bilirubin ≤ ULN; creatinine ≤ 1.5 mg/dL.
* If female of childbearing potential, pregnancy test is negative within 72 hours of first dose of study drug.
* If fertile, the patient agrees to use an effective method to avoid pregnancy for the duration of the study.
* Informed consent has been obtained.

Exclusion Criteria:

* Prior neo-adjuvant or adjuvant chemotherapy is allowed, and patients must have recovered from the acute toxicity of such therapies. No prior therapy for metastatic disease is allowed. If a taxane was part of the adjuvant regimen, at least 12 months should have passed from completion of taxane regimen to relapse. If a non-taxane-based adjuvant therapy was administered, at least 6 months should have passed from completion to relapse.
* Concurrent immunotherapy or hormonal therapy.
* Parenchymal brain metastases, including leptomeningeal involvement.
* Inadequately controlled hypertension (defined as blood pressure of > 150/100 mmHg) or New York Heart Association (NYHA) Grade 2 or greater congestive heart failure.
* Any prior history of hypertensive crisis or hypertensive encephalopathy.
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment.
* History of stroke or transient ischemic attack within 6 months prior to study enrollment.
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection).
* Symptomatic peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* History of abdominal fistula, gastrointestinal perforation, or intra- abdominal abscess within 6 months prior to study enrollment.
* Proteinuria at screening as demonstrated by either: - Urine protein:creatinine (UPC) ratio > 1.0 at screening OR - Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Known hypersensitivity to any component of bevacizumab.
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to first dose.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to first dose, anticipation of need for major surgical procedure during the course of the study. Serious, non-healing wound, ulcer, or bone fracture. Serious intercurrent medical or psychiatric illness, including serious active infection.
* History of other malignancy within the last 5 years which could affect the diagnosis or assessment of breast cancer.
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study.
* Pregnant or nursing women.
* Sensory neuropathy of > Grade 1 at baseline.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2010-07-01 (Actual); Study Completion 2011-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seidman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (40):
- United States (39):
  - Division of Hematology/Oncology University of Alabama at Birmingham, Birmingham, Alabama
  - Little Rock Hematology Oncology Associates, Little Rock, Arkansas
  - California Oncology of the Central Valley, Fresno, California
  - Glendale Memorial Hospital & Health Center, Glendale, California
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Oncology Associates of Bridgeport, Bridgeport, Connecticut
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Memorial Cancer Institute/Breast Cancer Center, Hollywood, Florida
  - Florida Cancer Institute, Hudson, Florida
  - Hematology Oncology Associates, Lake Worth, Florida
  - Medical Specialist of the Palm Beaches, Inc, Lake Worth, Florida
  - Gulfcoast Oncology Associates, St. Petersburg, Florida
  - Peachtree Hematology & Oncology Associates, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, PC, Marietta, Georgia
  - Center of Hope for Cancers and Blood, Stockbridge, Georgia
  - Maine Center for Cancer Medicine & Blood Disorders, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Harbor View Cancer Center, Baltimore, Maryland
  - Boston Medical Center Moakley Building, Solomont Center for Hematology & Medical Oncology, Boston, Massachusetts
  - North Shore Medical Cancer Center, Peabody, Massachusetts
  - St. John's Mercy Medical Center, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Drs. Forte, Schleidere, & Attas, PA, Englewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rosewell Park Cancer Institute Elm & Carlton Carlton Building, Buffalo, New York
  - Beth Israel Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Medical Oncology Aultman Hospital, Canton, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - Abington Hematology Oncology, Willow Grove, Pennsylvania
  - Family Cancer Center, Collierville, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - TX Oncology, PA, Austin, Texas
  - South Texas Oncology & Hematology Clinical Research Dept., San Antonio, Texas
  - Virginia Commonwealth University Medical Oncology, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Metropolitan Oncology Center, San Juan, Puerto Rico

REFERENCES:
- [Background] Seidman AD, Conlin AK, Bach A, Moynahan ME, Lake D, Forero A, Wright GS, Hackney MH, Clawson A, Norton L, Hudis CA. Randomized phase II trial of weekly vs. every 2 weeks vs. every 3 weeks nanoparticle albumin-bound paclitaxel with bevacizumab as first-line chemotherapy for metastatic breast cancer. Clin Breast Cancer. 2013 Aug;13(4):239-246.e1. doi: 10.1016/j.clbc.2013.02.008. PMID 23829890
- [Result] Conlin AK, Seidman AD, Bach A, Lake D, Dickler M, D'Andrea G, Traina T, Danso M, Brufsky AM, Saleh M, Clawson A, Hudis CA. Phase II trial of weekly nanoparticle albumin-bound paclitaxel with carboplatin and trastuzumab as first-line therapy for women with HER2-overexpressing metastatic breast cancer. Clin Breast Cancer. 2010 Aug 1;10(4):281-7. doi: 10.3816/CBC.2010.n.036. PMID 20705560

RESULTS

PARTICIPANT FLOW:
Groups:
- 260 mg/m^2 ABI-007 Every 3 Weeks: 260 mg/m^2 of ABI-007 every 3 weeks and 15 mg/kg bevacizumab every 3 weeks.
- 260 mg/m^2 ABI-007 Every 2 Weeks: 260 mg/m^2 of ABI-007 every two weeks and 10 mg/kg bevacizumab every 2 weeks
- 130 mg/m^2 ABI-007 Weekly: 130 mg/m^2 of ABI-007 every week and 10 mg/kg bevacizumab every 2 weeks
Period: Overall Study
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Started | 75 | 54 | 79
Completed | 0 (No participants completed because they continued in the study until disease progression) | 0 (No participants completed because they continued in the study until disease progression) | 0 (No participants completed because they continued in the study until disease progression)
Not Completed | 75 | 54 | 79
Not completed — Progressive Disease | 28 | 18 | 27
Not completed — Unacceptable Toxicity-related to trt | 21 | 24 | 32
Not completed — Adverse Event-unrelated to treatment | 3 | 0 | 2
Not completed — Physician Decision | 11 | 4 | 5
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 5 | 7
Not completed — Other | 6 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly | Total
Number analyzed (Participants) | 75 | 54 | 79 | 208
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 41 | 63 | 157
  >=65 years | 22 | 13 | 16 | 51
Age, Customized [Median (Full Range); unit: Years] | 59.0 [29.0 to 80.0] | 56.0 [36.0 to 79.0] | 56.0 [32.0 to 85.0] | 57.0 [29.0 to 85.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 54 | 79 | 208
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1 | 2
  Black, of African Heritage | 11 | 13 | 19 | 43
  White, Non-Hispanic and Non-Latino | 52 | 31 | 45 | 128
  White, Hispanic or Latino | 8 | 10 | 14 | 32
  Other (not specified) | 3 | 0 | 0 | 3
Weight [Median (Full Range); unit: kilograms] | 72.9 [41.8 to 119.5] | 70.2 [41.4 to 145.0] | 73.1 [46.0 to 167.8] | 72.2 [41.4 to 167.8]
Menopausal status [Number; unit: Participants]
  Pre-menopausal | 11 | 11 | 16 | 38
  Post-menopausal | 64 | 43 | 63 | 170
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    0 | 43 | 33 | 48 | 124
    1 | 29 | 17 | 27 | 73
    2 | 3 | 4 | 4 | 11
    3 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0
Time from Primary Diagnosis to Study Entry [Median (Full Range); unit: Years] | 4.320 [0.025 to 16.901] | 3.127 [0.041 to 23.932] | 2.579 [0.022 to 21.065] | 2.983 [0.022 to 23.932]
Participants with Current Diagnosis at Stage IV [Number; unit: Participants] — Stage IV characteristics are the cancer can be any size (any T) and may or may not have spread to nearby lymph nodes (any N). It has spread to distant organs or to lymph nodes far from the breast (M1). The most common sites of spread are the bone, liver, brain, or lung,
  Participants | 75 | 54 | 79 | 208

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Confirmed Complete Response (CR) or Partial Response (PR) Based on Response Evaluation Criteria In Solid Tumors (RECIST v1.0)
Description: Using the RECIST response criteria version 1.0, the percent of participants achieving either a complete response (CR) defined as the disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation or partial response (PR) defined as at least a 30% decrease in the sum of the longest diameters of target lesions and no progression in non-target lesions based on confirmed responses from the investigator assessment of best overall response during study treatment.
Time Frame: Up to 43 months
Population: Treated population
Measure: Number; unit: Percent of Total Participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Percent of Total Participants | 41 | 43 | 47
Statistical Analysis 1: Comparison: 260 mg/m^2 ABI-007 Every 3 Weeks vs 130 mg/m^2 ABI-007 Weekly; Test type: Superiority or Other; p = 0.4476, Cochran-Mantel-Haenszel — Group comparison was performed between group 260 mg/m^2 ABI-007 every 3 weeks and group 130 mg/m^2 ABI-007 weekly, as based on amended protocol, no type I error adjustment for multiplicity; a priori threshold for statistical significance is 0.05; Stratified by study site

2. Secondary Outcome: Percentage of Participants With Stable Disease for ≥ 16 Weeks, or Complete or Partial Overall Response (i.e., Total Response) Based on Response Evaluation Criteria In Solid Tumors (RECIST v1.0)
Description: Using Response Evaluation Criteria in Solid Tumors (RECIST v1.0), the percentage of participants achieving either
  * A complete response (CR) defined as the disappearance of all known disease and no new sites or disease related symptoms confirmed at least 4 weeks after initial documentation or
  * A partial response (PR) defined as at least a 30% decrease in the sum of the longest diameters of target lesions and no progression in non-target lesions or
  * Stable disease (SD) defined as neither sufficient shrinkage to qualify for PR or sufficient increase to qualify for progressive disease.
Time Frame: Up to 43 months (until progressed)
Population: Treated population
Measure: Number; unit: Percent of Total Participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Percent of Total Participants | 65 | 52 | 58

3. Primary Outcome: Participant Counts of the Most Severe Grade for Absolute Neutrophil (ANC) as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Experience (NCI CTCAE v3)
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest measured (nadir) ANC counts were graded using NCI CTCAE version 3:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 75.0*10^9L; Grade 2 = <1.5 - 1.0*10^9L; Grade 3 = <1.0 - 0.5*10^9L; Grade 4 = <0.5*10^9L
Time Frame: up to 54 months
Population: Treated population who had at least one post baseline value
Measure: Number; unit: participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 63 | 49 | 70
participants
  Grade 0 | 51 (1.569) | 34 (3.216) | 17 (.750)
  Grade 1 | 5 | 5 | 17
  Grade 2 | 2 | 6 | 17
  Grade 3 | 3 | 4 | 17
  Grade 4 | 2 | 0 | 2

4. Secondary Outcome: Kaplan Meier Estimate for Time to Disease Progression (TTP)
Description: Time to progression was defined as the time from the first dose of study drug to the start of progression. Participants that did not have progression were censored at the last known time the patient was evaluated for progression. Participants that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
  Progressive disease was defined as at least a 20% increase in the sum of the longest diameters of target lesions; or the appearance of one or more new lesions; or the unequivocal progression of a non-target lesion.
Time Frame: Up to 43 months (until progressed)
Population: Treated population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Months | 8.0 [7.0 to 10.3] | 6.3 [5.3 to 8.0] | 9.0 [7.2 to 11.1]

5. Secondary Outcome: Kaplan Meier Estimate for Duration of Response
Description: Duration of response was defined as the time from response to the time of disease progression for participants who achieve an objective confirmed complete (CR) or partial overall response (PR). Disease progression is based on the assessments by the investigator. Participants who did not have disease progression following a confirmed complete or partial target response were censored at the last known time that the participant was evaluated for response
Time Frame: Up to 43 months (until progressed)
Population: Treated population who achieved a complete or partial response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 33 | 22 | 36
Months | 10.3 [8.0 to 12.3] | 8.0 [5.5 to 13.4] | 9.9 [7.7 to 15.7]

6. Secondary Outcome: Kaplan Meier Estimate for Participant Survival
Description: Participant survival was summarized using Kaplan-Meier estimate of the time of first dose of study drug to the last known time that the participant was alive. Participants that were alive at the end of follow-up would be censored at the last known time that the patient was alive.
Time Frame: Up to 56 months
Population: Treated population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Months | 21.3 [19.5 to 26.6] | 19.0 [15.0 to 28.1] | 23.7 [18.2 to 31.0]

7. Primary Outcome: Participant Counts of the Most Severe Grade for White Blood Cells (WBC) as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Experience (NCI CTCAE v3)
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest measured (nadir) WBC counts were graded using NCI CTCAE version 3:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal -3.0*10^9/L; Grade 2 = <3.0 - 2.0*10^9/L; Grade 3 = <2.0 - 1.0*10^9/L; Grade 4 = <1.0*10^9/L
Time Frame: up to 54 months
Population: Treated population who had at least one post baseline value
Measure: Number; unit: participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 64 | 49 | 70
participants
  Grade 0 | 47 | 30 | 11
  Grade 1 | 9 | 14 | 21
  Grade 2 | 6 | 5 | 26
  Grade 3 | 2 | 0 | 11
  Grade 4 | 0 | 0 | 1

8. Primary Outcome: Participant Counts of the Most Severe Grade for Platelet Counts as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Experience (NCI CTCAE v3)
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest measured (nadir) platelet counts were graded using NCI CTCAE version 3:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 75.0*10^9/L; Grade 2 = <75.0 - 50.0*10^9/L; Grade 3 = <50.0 - 25.0*10^9/L; Grade 4 = <25.0*10^9/L
Time Frame: up to 54 months
Population: Treated population who had at least one post baseline value
Measure: Number; unit: participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 63 | 49 | 70
participants
  Grade 0 | 60 | 39 | 64
  Grade 1 | 2 | 10 | 4
  Grade 2 | 1 | 0 | 1
  Grade 3 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0

9. Primary Outcome: Participant Counts of the Most Severe Grade for Hemoglobin Levels as Graded by the National Cancer Institute Common Terminology Criteria for Adverse Experience (NCI CTCAE v3)
Description: Myelosuppression is a decrease in the ability of the bone marrow to produce blood cells. The lowest measured (nadir) hemoglobin levels were graded using NCI CTCAE version 3:
  Grade 0 = within normal limits; Grade 1 = < lower limit of normal - 100g/L; Grade 2 = <100 - 80g/L; Grade 3 = <80 - 65g/L; Grade 4 = <65g/L
Time Frame: up to 54 months
Population: Treated population who had at least one post baseline value
Measure: Number; unit: participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 64 | 49 | 70
participants
  Grade 0 | 41 | 25 | 13
  Grade 1 | 17 | 18 | 33
  Grade 2 | 6 | 6 | 19
  Grade 3 | 0 | 0 | 4
  Grade 4 | 0 | 0 | 1

10. Primary Outcome: The Number of Participants With at Least One Dose Reduction for ABI-007
Description: Participants with at least one dose reduction for ABI-007. ABI-007 (Abraxane) dose could be reduced according to protocol guidelines if the participant was experiencing toxicities. Participants were allowed two ABI-007 (Abraxane) dose reductions during the course of the trial. This outcome is considered to be both a safety and an efficacy outcome.
Time Frame: Up to 53 months
Population: Treated population
Measure: Number; unit: Participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Participants | 36 | 32 | 53

11. Primary Outcome: The Number of Participants With at Least One Dose Delay for ABI-007
Description: Participants with at least one dose delay for ABI-007. Treatment delays of no longer than 2 weeks allowed participants to recovery from acute toxicity. If treatment was delayed beyond 2 weeks, continuing treatment on protocol was at the physician's discretion, based upon the best interests of the participant. This outcome is considered to be both a safety and an efficacy outcome.
Time Frame: Up to 53 months
Population: Treated population
Measure: Number; unit: Participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Participants | 40 | 27 | 68

12. Primary Outcome: The Number of Participants With a Dose Interruption of ABI-007
Description: Number of participants who interrupted (omitted) a dose at some point in the treatment period. This outcome is considered to be both a safety and an efficacy outcome.
Time Frame: Up to 53 months
Population: Treated population
Measure: Number; unit: Participants
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
Participants | 2 | 0 | 0

13. Secondary Outcome: Kaplan Meier Estimate for Progression-Free Survival (PFS)
Description: PFS was defined as the time from the first dose of study drug to the start of progression or patient death (any cause) whichever occurred first. Participants that did not have progression or have not died were censored at the last known time the participant was progression free. Participants that initiate other anticancer therapy prior to progression were censored at the time when new anticancer therapy was initiated.
Time Frame: up to 56 months
Population: Treated population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Number analyzed (Participants) | 75 | 54 | 79
months | 7.7 [7.3 to 8.8] | 6.3 [5.3 to 8.0] | 8.8 [5.8 to 9.9]

ADVERSE EVENTS:
Time Frame: Up to 54 months
Arm/Group | 260 mg/m^2 ABI-007 Every 3 Weeks | 260 mg/m^2 ABI-007 Every 2 Weeks | 130 mg/m^2 ABI-007 Weekly
Serious Adverse Events (participants affected / at risk) | 22/75 | 16/54 | 32/79
Other Adverse Events (participants affected / at risk) | 75/75 | 54/54 | 78/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 260 mg/m^2 ABI-007 Every 3 Weeks (N=75) | 260 mg/m^2 ABI-007 Every 2 Weeks (N=54) | 130 mg/m^2 ABI-007 Weekly (N=79)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (2)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Breast cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 5 (5)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cranial neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 260 mg/m^2 ABI-007 Every 3 Weeks (N=75) | 260 mg/m^2 ABI-007 Every 2 Weeks (N=54) | 130 mg/m^2 ABI-007 Weekly (N=79)
Anaemia (Blood and lymphatic system disorders) | 15 (24) | 20 (32) | 24 (37)
Leukopenia (Blood and lymphatic system disorders) | 6 (32) | 4 (7) | 11 (23)
Neutropenia (Blood and lymphatic system disorders) | 18 (52) | 9 (13) | 31 (63)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 5 (5)
Dry eye (Eye disorders) | 5 (5) | 0 (0) | 4 (6)
Lacrimation increased (Eye disorders) | 3 (3) | 5 (5) | 14 (22)
Vision blurred (Eye disorders) | 9 (10) | 9 (10) | 11 (13)
Visual disturbance (Eye disorders) | 4 (5) | 1 (2) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 3 (5) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 9 (16) | 2 (2) | 11 (12)
Abdominal pain upper (Gastrointestinal disorders) | 4 (6) | 1 (1) | 9 (10)
Constipation (Gastrointestinal disorders) | 30 (41) | 28 (29) | 38 (54)
Diarrhoea (Gastrointestinal disorders) | 24 (42) | 24 (36) | 43 (62)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 3 (4) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 11 (13) | 2 (3) | 6 (6)
Dysphagia (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 8 (8)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (2) | 5 (5)
Haemorrhoids (Gastrointestinal disorders) | 3 (3) | 2 (2) | 6 (6)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (3)
Nausea (Gastrointestinal disorders) | 37 (53) | 36 (53) | 40 (58)
Oral pain (Gastrointestinal disorders) | 1 (1) | 4 (4) | 4 (5)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 6 (7)
Stomatitis (Gastrointestinal disorders) | 10 (14) | 8 (9) | 13 (18)
Vomiting (Gastrointestinal disorders) | 16 (20) | 18 (25) | 21 (28)
Asthenia (General disorders) | 4 (5) | 11 (13) | 8 (10)
Chest pain (General disorders) | 2 (2) | 4 (5) | 7 (9)
Chills (General disorders) | 6 (8) | 4 (4) | 11 (13)
Fatigue (General disorders) | 55 (127) | 43 (82) | 64 (137)
Gait disturbance (General disorders) | 1 (1) | 2 (2) | 4 (4)
Mucosal inflammation (General disorders) | 14 (17) | 13 (15) | 16 (28)
Oedema (Gastrointestinal disorders) | 1 (1) | 1 (1) | 5 (6)
Oedema peripheral (General disorders) | 6 (10) | 10 (11) | 11 (15)
Pain (General disorders) | 6 (6) | 11 (13) | 11 (15)
Pyrexia (General disorders) | 9 (10) | 11 (12) | 11 (19)
Hypersensitivity (Immune system disorders) | 1 (1) | 3 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (8)
Nail infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (5)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 5 (7)
Oral candidiasis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Sinusitis (Infections and infestations) | 4 (4) | 3 (3) | 7 (9)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 5 (5) | 9 (9)
Urinary tract infection (Infections and infestations) | 13 (21) | 9 (10) | 12 (13)
Haemoglobin decreased (Investigations) | 2 (2) | 3 (3) | 3 (4)
Weight decreased (Investigations) | 4 (7) | 9 (11) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 16 (20) | 19 (26) | 24 (33)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 4 (4) | 6 (6)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 7 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 (60) | 21 (24) | 16 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 9 (10) | 11 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (16) | 18 (22) | 6 (9)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4) | 5 (5) | 7 (7)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (14) | 10 (14) | 10 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 (20) | 11 (16) | 14 (19)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 6 (8)
Coordination abnormal (Nervous system disorders) | 5 (5) | 1 (4) | 3 (3)
Dizziness (Nervous system disorders) | 15 (17) | 10 (10) | 11 (13)
Dysgeusia (Nervous system disorders) | 14 (16) | 14 (17) | 28 (36)
Headache (Nervous system disorders) | 15 (17) | 11 (14) | 18 (28)
Hypoaesthesia (Nervous system disorders) | 1 (3) | 3 (5) | 4 (4)
Neuropathy (Nervous system disorders) | 34 (96) | 24 (77) | 34 (94)
Neuropathy peripheral (Nervous system disorders) | 15 (36) | 9 (12) | 13 (41)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 3 (4) | 4 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 34 (104) | 24 (63) | 36 (111)
Anxiety (Psychiatric disorders) | 4 (4) | 7 (7) | 8 (8)
Depression (Psychiatric disorders) | 12 (12) | 8 (9) | 11 (13)
Insomnia (Psychiatric disorders) | 17 (19) | 17 (18) | 10 (11)
Dysuria (Renal and urinary disorders) | 5 (5) | 4 (4) | 2 (4)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 4 (5)
Proteinuria (Renal and urinary disorders) | 5 (5) | 1 (1) | 3 (4)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 8 (9) | 20 (26)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 9 (11) | 21 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 32 (44) | 23 (25) | 42 (53)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 8 (10) | 8 (9)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 4 (4) | 4 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 9 (11)
Alopecia (Skin and subcutaneous tissue disorders) | 49 (51) | 35 (45) | 53 (68)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 8 (8) | 12 (12)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 5 (6)
Nail discolouration (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (6) | 10 (11)
Nail disorder (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (11) | 23 (42)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5) | 2 (2)
Onychorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 3 (4) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 20 (23) | 17 (25) | 31 (42)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 7 (8)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2) | 3 (3) | 4 (4)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 7 (9)
Hot flush (Vascular disorders) | 5 (7) | 4 (5) | 7 (7)
Hypertension (Vascular disorders) | 19 (27) | 9 (9) | 11 (17)
Lymphoedema (Vascular disorders) | 1 (1) | 1 (1) | 8 (12)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4)
Blood pressure increased (Investigations) | 4 (4) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Upon investigator submission of a publication or presentation to Celgene, Celgene shall complete its review within 60 days after receipt of the proposed publication or presentation. Upon Celgene's request, proposed publication or presentation will be delayed up to 60 additional days to enable Celgene to secure adequate intellectual property protection of property of Celgene that would be affected by such proposed publication or presentation